CLINICAL TRIAL: NCT03455426
Title: Intrauterine Insemination With Letrozole Versus Intrauterine Insemination in Natural Cycle. A Randomised Controlled Trial
Brief Title: Intrauterine Insemination With Letrozole Versus in Natural Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jie Qiao, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUI-letrozole/natural cycle
Record Dates: First submitted 2018-02-25; First posted 2018-03-06 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2019-07

CONDITIONS: Infertility; Intrauterine Insemination
MeSH Terms: conditions — Infertility | interventions — Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- letrozole group (Experimental): letrozole 5mg/day starting from day 3 of menstrual cycle for 5 days
  Interventions: Drug: letrozole
- natural cycle group (No Intervention)

INTERVENTIONS:
Drug: letrozole — Women will be randomizedfor ovarian stimulation with letrozole or to natural cycle IUI.
  Arms: letrozole group

SUMMARY:
Rationale: Intrauterine insemination (IUI) is the treatment of first choice for couples with unexplained and mild male factor infertility in many countries, but it is controversial whether ovarian stimulation improves fertility outcomes. In recent retrospectively collected data, investigators found that in couples with unexplained and mild male factor infertility undergoing IUI, ovarian stimulation with letrozole increased live birth rate as compared to natural cycle IUI without substantially increasing the multiple pregnancy rate. Investigators therefore perform a randomized clinical trial (RCT) on the subject in the Centre of Reproductive Medicine, Peking University Third Hospital, Beijing, China.

Objective: To test the hypothesis that in couples with unexplained or mild male factor infertility scheduled for an IUI program ovarian stimulation with letrozole increases the live birth rate as compared to natural cycle treatment.

Study design Randomized clinical trial.

Study population Women diagnosed with unexplained or mild male factor infertility scheduled for treatment with IUI.

Intervention Women will be randomized for ovarian stimulation with letrozole or to natural cycle IUI. In the group allocated to ovarian stimulation, women will receive oral tablets letrozole 5 mg daily from cycle day 3-5 for 5 days. Investigators will treat the couples for 3 cycles, with a time horizon of 4 months.

Main study parameters/endpoints Primary outcome is ongoing pregnancy leading to live birth. Secondary endpoints are clinical pregnancy, multiple pregnancy, miscarriage rates, pregnancy complications and patients' costs.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness The strategies compared are already broadly applied in current practice. No additional risks are expected. There is no benefit for participants, but the results may benefit future subfertile couples.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with unexplained or mild male subfertility
* At least one sided tubal patency, established according to local protocol
* Normal or mild impairment of semen quality defined as a TMSC of 3 million or more based on at least one semen analysis

Exclusion Criteria:

* Woman with double sided tubal pathology
* Women with irregular cycles, PCOS or other endocrine disorders
* Impaired semen quality: pre-wash TMSC <3 million.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy | 3 months
  Primary outcome is ongoing pregnancy leading to live birth

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Huang, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Franik S, Le QK, Kremer JA, Kiesel L, Farquhar C. Aromatase inhibitors (letrozole) for ovulation induction in infertile women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2022 Sep 27;9(9):CD010287. doi: 10.1002/14651858.CD010287.pub4. PMID 36165742

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT03455426/Prot_SAP_000.pdf